CLINICAL TRIAL: NCT00460226
Title: A Multi-centre, Observational Study to Evaluate the Incidence of Non-serious Rash in Korean Bipolar I Patients With Lamotrigine Therapy in Real World Setting
Brief Title: Lamictal Bipolar Observational Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: LBI108245
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorder
Keywords: Korean; Bipolar I disorder; Non-serious rash; Lamotrigine
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- lamotrigine: there is only one group.
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine — lamotrigine treatment for 12weeks

SUMMARY:
This is multi-center, prospective, observational stud. This study is designed to evaluate the rate of non-serious rash in Korean bipolar I patients.

ELIGIBILITY:
Inclusion criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Provides written informed consent
* Male or female age 18 years or older A female subject is eligible to enter and participate in the study if she is of;
* Non-childbearing potential
* Childbearing potential, has a negative pregnancy test at screen
* Diagnosis of bipolar I disorder using DSM-IV criteria

Exclusion criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Previous or current treatment with lamotrigine
* Presence of a clinically significant psychiatric or physiologic comorbidity, including significant substance abuse, severe depression or mania which is of an unstable or progressive nature that could, in the opinion of the investigator, interfere with participation in this study
* Presence of untreated thyroid disease
* Have active suicidality or homicidality, history of recent suicide attempts within the past year, or, in the investigator's opinion, a marked risk for suicide
* History of severe hepatic or renal insufficiency or significant hematologic disease or other significant medical or psychiatric condition that would interfere with subjects' participation in the study
* Currently participating in another clinical trial, or plans to enroll in another trial while participating in this study
* Currently pregnant or is breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient setting and reflecting usual clinical practice in general hospital
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of non-serious rash during 12 weeks of treatment with lamotrigine in patients with bipolar I in Korea | 12 weeks

SECONDARY OUTCOMES:
CGI-BP at Week 12 and occurrence of adverse events at Week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Woo YS, Bahk WM, Jon DI, Joo YH, Kim W, Seo JS, Ahn YM, Chung SK, Won SH, Shin YC, Yoon BH, Jung SH, Seok JH, Lee YS, Kim Y, Min KJ. Rash in adult patients receiving lamotrigine to treat bipolar I disorder in Korea: a multicenter, prospective, naturalistic, open-label trial. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Oct 1;33(7):1147-52. doi: 10.1016/j.pnpbp.2009.06.010. Epub 2009 Jun 18. PMID 19540298